CLINICAL TRIAL: NCT05967741
Title: Randomized Controlled Clinical Trial to Gauge the Effects of Dietary Erythritol on Platelet Reactivity and Vascular Inflammation
Brief Title: The Effects of Dietary Erythritol on Platelet Reactivity and Vascular Inflammation
Acronym: EASI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2030510
Record Dates: First submitted 2023-06-06; First posted 2023-08-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Platelet Aggregation, Spontaneous; Vascular Thrombosis
Keywords: platelet activation; vascular inflammation; erythritol; aspartame; dietary intervention
MeSH Terms: conditions — Platelet Aggregation, Spontaneous; Thrombosis | interventions — Erythritol; Ethanol; Aspartame

STUDY DESIGN:
Intervention Model Description: Randomized crossover study with 2-week washout
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Experimental and control beverage are formulated to be similar color, taste and volume.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythritol-sweetened beverage (Experimental): 1-gram erythritol/kg body weight/day, divided into three beverage servings and fruit-flavored with Kool-Aid® unsweetened drink mix.
  Interventions: Other: Erythritol
- Aspartame-sweetened beverage (Placebo Comparator): Control beverages will be made from a noncaloric aspartame-sweetened, fruit-flavored drink mix at the concentration needed to match the sweetness (~3 mg aspartame/kg/day) and flavoring of the erythritol beverages on a per volume basis.
  Interventions: Other: Aspartame

INTERVENTIONS:
Other: Erythritol — Erythritol is a naturally occurring and non-nutritive sugar alcohol that is classified as generally recognized as safe (GRAS)
  Other Names: Noncaloric sugar alcohol
  Arms: Erythritol-sweetened beverage
Other: Aspartame — Aspartame consists of two amino acids, phenylalanine and aspartic acid, and a methyl group. It does not have metabolic effects and has served as the blinded control beverage in the investigators' completed NIH-funded clinical trials.
  Other Names: Noncaloric sweetener
  Arms: Aspartame-sweetened beverage

SUMMARY:
The purpose is to conduct a dietary intervention study in which human participants will consume beverages sweetened with erythritol or aspartame, each for 2 weeks, in a randomized crossover design

DETAILED DESCRIPTION:
There is a strong correlation between plasma erythritol concentrations and adverse cardiovascular events in high risk individuals. It has also been demonstrated that consumption of dietary erythritol leads to high levels of plasma erythritol. There is in vitro evidence that erythritol at comparable concentrations promotes platelet activation. However, there is no direct evidence that links human consumption of erythritol with the onset of platelet activation and adhesion leading to inflammation. The investigators seek to fill this evidence gap by conducting a randomized crossover dietary intervention study in which human participants will consume beverages sweetened with erythritol or aspartame, each for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27 kg/m2

Exclusion Criteria:

* • History of blood clot, transient ischemic attack (TIA), stroke, angina, heart attack, or peripheral vascular disease, or current cancer diagnosis.

  * Pregnant or lactating women
  * Current, prior (within 12 months), or anticipated use of medications for treatment of hyperlipidemia, high blood pressure or diabetes, or any medication that in the opinion of the investigators will confound results.
  * Unwilling to forego the use of anti-inflammatory medication during study.
  * Unwilling to forego the use of marijuana during the study.
  * Use of tobacco.
  * Strenuous exerciser (>4 hours/week at a level more vigorous than walking).
  * Surgery or medication for weight loss.
  * Diet exclusions: Food allergies or dietary restrictions that may undermine compliance to dietary protocol, routine ingestion of more than 2 sugar-sweetened beverages or 2 alcoholic beverage/day. Unwillingness to consume artificial or noncaloric sweeteners. Habitual consumption (>10 gram/day) of beverage or foods that contain erythritol. Recent or current weight loss diet.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
P-selectin, a platelet surface marker, assessed as median fluorescence intensity | 6 weeks
  Change in median fluorescence intensity of P-selectin, an index of platelet activation, will be measured by flow cytometry in whole blood collected from subjects before and after consuming erythritol-sweetened beverage for 2 weeks and compared with change in whole blood collected before and after consuming aspartame-sweetened beverage for 2 weeks
P-selectin, a platelet surface marker, assessed as percentage of P-selectin positive cells | 6 weeks
  Change in percentage of P-selectin positive cells, an index of platelet activation, will be measured by flow cytometry in whole blood collected from subjects before and after consuming erythritol-sweetened beverage for 2 weeks and compared with change in whole blood collected before and after consuming aspartame-sweetened beverage for 2 weeks
PAC-1 (GPIIb/IIIa complex), a platelet surface marker, assessed as median fluorescence intensity | 6 weeks
  Change in median fluorescence intensity of PAC-1, an index of platelet activation, will be measured by flow cytometry in whole blood collected from subjects before and after consuming erythritol-sweetened beverage for 2 weeks and compared with change in whole blood collected before and after consuming aspartame-sweetened beverage for 2 weeks
PAC-1 (GPIIb/IIIa complex), a platelet surface marker, assessed as percentage of PAC-1 positive cells | 6 weeks
  Change in percentage of PAC-1 positive cells, an index of platelet activation, will be measured by flow cytometry in whole blood collected from subjects before and after consuming erythritol-sweetened beverage for 2 weeks and compared with change in whole blood collected before and after consuming aspartame-sweetened beverage for 2 weeks
Annexin V, a platelet surface marker, assessed as median fluorescence intensity | 6 weeks
  Change in median fluorescence intensity of annexin V, an index of platelet activation, will be measured by flow cytometry in whole blood collected from subjects before and after consuming erythritol-sweetened beverage for 2 weeks and compared with change in whole blood collected before and after consuming aspartame-sweetened beverage for 2 weeks
Annexin V, a platelet surface marker, assessed as percentage of annexin V positive cells | 6 weeks
  Change in percentage of annexin V positive cells, an index of platelet activation, will be measured by flow cytometry in whole blood collected from subjects before and after consuming erythritol-sweetened beverage for 2 weeks and compared with change in whole blood collected before and after consuming aspartame-sweetened beverage for 2 weeks
Platelet reactivity to physiologic agonist, assessed as change in median fluorescence intensity | 6 weeks
  The change in median fluorescence intensity induced by physiologic agonists, an index of platelet reactivity, will be measured by flow cytometry in whole blood collected from subjects before and after consuming erythritol-sweetened beverage for 2 weeks and compared with change in whole blood collected before and after consuming aspartame-sweetened beverage for 2 weeks
Platelet aggregation in response to physiologic agonist, assessed as aggregation/min | 6 weeks
  The change in aggregation/min induced by physiologic agonists will be measured by light transmission aggregometry in whole blood collected from subjects before and after consuming erythritol-sweetened beverage for 2 weeks and compared with change in whole blood collected before and after consuming aspartame-sweetened beverage for 2 weeks
Platelet aggregation in response to physiologic agonist, assessed as percent of maximum aggregation | 6 weeks
  The change in % maximum aggregation induced by physiologic agonists will be measured by light transmission aggregometry in whole blood collected from subjects before and after consuming erythritol-sweetened beverage for 2 weeks and compared with change in whole blood collected before and after consuming aspartame-sweetened beverage for 2 weeks
Platelet-leukocyte interaction, assessed as platelet/leukocyte aggregate size by fluorescence mean intensity | 6 weeks
  Change in platelet/leukocyte aggregate size, an index of platelet-leukocyte interaction, will be measured by flow cytometry in whole blood collected from subjects before and after consuming erythritol-sweetened beverage for 2 weeks and compared with change in whole blood collected before and after consuming aspartame-sweetened beverage for 2 weeks

SECONDARY OUTCOMES:
Plasma concentration of E-Selectin | 6 weeks
  Change in plasma E-Selectin in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of sVCAM1 | 6 weeks
  Change in plasma sVCAM1 in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of sICAM1 | 6 weeks
  Change in plasma sICAM1 in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of D-dimer | 6 weeks
  Change in plasma D-dimer in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of Platelet factor 4 | 6 weeks
  Change in plasma platelet factor 4 in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of Fibrinogen | 6 weeks
  Change in plasma fibrinogen in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of Prothrombin fragment 1+2 | 6 weeks
  Change in plasma prothrombin fragment 1+2 in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of Plasmin-antiplasmin complex | 6 weeks
  Change in plasma plasmin-antiplasmin complex in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of Lp(a) | 6 weeks
  Change in plasma Lp(a) in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage

OTHER OUTCOMES:
Plasma concentration of glucose | 6 weeks
  Change in plasma fasting glucose in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of triglyceride | 6 weeks
  Change in plasma fasting triglyceride in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of cholesterol | 6 weeks
  Change in plasma fasting cholesterol in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of low density lipoprotein cholesterol | 6 weeks
  Change in plasma fasting low density lipoprotein cholesterol in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of high density lipoprotein cholesterol | 6 weeks
  Change in plasma fasting high density lipoprotein cholesterol in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of apolipoprotein B | 6 weeks
  Change in plasma fasting apolipoprotein B in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of apolipoprotein CIII | 6 weeks
  Change in plasma fasting apolipoprotein CIII in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage
Plasma concentration of uric acid | 6 weeks
  Change in plasma fasting uric acid in subjects before and after sustained consumption of erythritol-sweetened beverage compared with change before and after sustained consumption of aspartame-sweetened beverage

CONTACTS AND LOCATIONS:
Locations (1):
- Ragle Human Nutrition Research Center, University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Witkowski M, Nemet I, Alamri H, Wilcox J, Gupta N, Nimer N, Haghikia A, Li XS, Wu Y, Saha PP, Demuth I, Konig M, Steinhagen-Thiessen E, Cajka T, Fiehn O, Landmesser U, Tang WHW, Hazen SL. The artificial sweetener erythritol and cardiovascular event risk. Nat Med. 2023 Mar;29(3):710-718. doi: 10.1038/s41591-023-02223-9. Epub 2023 Feb 27. PMID 36849732